CLINICAL TRIAL: NCT03902249
Title: Effect of Intravenous Dexamethasone in Combination With Pudendal Nerve Block on Postoperative Pain Control in Pediatric Hypospadias Repair
Brief Title: Effect of Intravenous Dexamethasone With Pudendal Nerve Block on Postoperative Pain in Pediatric Hypospadias Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Sonia ben khalifa (PhD) (Other)
Responsible Party: Sponsor-Investigator, Dr Sonia ben khalifa (PhD), Clinical Professor, Hôpital d'enfants Béchir-Hamza
Organization: Hôpital d'enfants Béchir-Hamza (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DexaProtocol
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain; Hypospadias
Keywords: Intravenous Dexamethasone; Pudendal nerve block; Analgesia; Postoperative pain; Children; Hypospadias
MeSH Terms: conditions — Pain, Postoperative; Hypospadias; Agnosia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Active Comparator): Patients who received 0.15mg/kg of Dexamethasone in 8ml of saline
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): Patients who received the same volume of saline as the study group (8ml)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
This study aims to determine if intravenous Dexamethasone combined with a pudendal nerve block is able to prolong postoperative analgesia in children undergoing hypospadias repair.

DETAILED DESCRIPTION:
It was a prospective study, randomized, double blind study, conducted at the Tunis Children's Hospital (January 2017-December 2018). After agreement with parents and the local ethics committee, the investigators included children aged 1 to 18 years, ASA 1-2, proposed for a hypospadias repair. Patients were randomized to: Group D receiving 0. 15mg/kg of Dexamethasone IV after induction and group P receiving the same volume of saline. The pudendal block was performed by neurostimulation after induction with Sevoflurane and 3 gamma/kg Fentanyl IV. The success of the block was tested at 10 and 15 minutes, it was declared successful when the systolic blood pressure and heart rate did not increase by more than 20% compared to the baseline values at the time of the incision. No analgesics were administered at the end of the surgery. The pain was assessed by the CHEOPS score the first 24 hours. The X2 test was used for qualitative variables and the student test for quantitative variables with P<0. 05 as the significance threshold. The number of patients required for the study was calculated (alpha=5% beta=90%) and was 62.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification 1 or 2
* Procedure: hypospadias repair
* Eligible for a pudendal nerve block

Exclusion Criteria:

* parents or patient refusal
* nerve block failure
* Peroperative complication.

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The mean time to first rescue analgesic | The first 24 hours after surgery
  Time from the end of surgery to the first administration of rescue analgesic
number of rescue analgesic consumption | The first 24 hours after surgery
  Total number of rescue analgesic consumption for each patient

SECONDARY OUTCOMES:
pain scores (CHEOPS) | Hour 0, Hour 1, Hour 2, Hour 3, Hour 4, Hour 8, Hour 12, Hour 24
  CHEOPS score ranges from 4 to 13. 13 is the worst score. If the score was superior to 7 rescue analgesia was administrated.
Number of episodes of postoperative nausea and vomiting | The first 24 hours after surgery
  Number of episodes of postoperative nausea and vomiting in each patient

REFERENCES:
- [Derived] Khalifa SB, Slimene AB, Blaiti H, Kaddour R, Hassen AF, Pardessus P, Brasher C, Dahmani S. The potentiating effect of intravenous dexamethasone upon preemptive pudendal block analgesia for hypospadias surgery in children managed with Snodgrass technique: a randomized controlled study : Dexamethasone for pain management in children. BMC Anesthesiol. 2024 Apr 16;24(1):145. doi: 10.1186/s12871-024-02536-3. PMID 38627668